CLINICAL TRIAL: NCT04413890
Title: Administration of Prostaglandin Gel for Cervical Priming During Induction of Labour Every 12 Hours Versus 24 Hours: a Randomized Superiority Controlled Trial
Brief Title: Comparison of Two Rhythm of Administration of Prostaglandin Gel for Induction of Labor
Acronym: GELFREQ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19_RIPH2_10
Record Dates: First submitted 2020-04-07; First posted 2020-06-04 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Labor Complication; Cervix
Keywords: Induction; Term; Labor; Rhythm; Prostaglandins
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical administration (Active Comparator): One prostaglandin vaginal gel every 24 hours
  Interventions: Drug: Dinoprostone vaginal gel
- Experimental administration (Experimental): One prostaglandin vaginal gel every 12 hours
  Interventions: Drug: Dinoprostone vaginal gel

INTERVENTIONS:
Drug: Dinoprostone vaginal gel — Prostaglandin gel 0.5, 1 or 2 mg
  Other Names: cervical priming with prostaglandin gel

SUMMARY:
The study compares two rhythms of administration of prostaglandin vaginal gels for cervical priming before induction of labor in term patients. In our institution, prostaglandin gels are given for a maximum of three times, with induction by oxytocin and amniotomy the day after the last gel whatever Bishop score has been obtained. This management results in some patient spending four days in hospital before delivery. The aim of the study is to compare our classical management scheme with a reduced interval between to gels, of 12h instead of 24 h. The primary outcome will be the time elapsed between the first prostaglandin gel and delivery. Tolerance of both management patterns will also be evaluated through a satisfaction survey.

DETAILED DESCRIPTION:
Approximatively 22% of pregnant women have an induction of labor in France (22.9% in our institution in 2019), mainly for prolonged pregnancy after 41 weeks gestational age or prolonged rupture of membranes. Patients whose cervix is considered unripe (Bishop score under 6) are generally proposed a cervical priming because induction of labor without prior priming entails a higher of cesarean delivery rate for failed induction. The devices used for cervical priming are pharmacological (mainly prostaglandin gel, pessaries or suppositories) or mechanical (Foley catheter, Cook balloons). Very few recommendations exist regarding the type of device, the rhythm and maximal number of repeat administrations and the interval between two administrations. Shortening interval between two administrations (in case of use of a device necessitating serial prescriptions) may shorten the time interval between beginning of priming and delivery. In our institution, a vaginal gel can be given three times before induction of labor with oxytocin and amniotomy, whatever Bishop score has been obtained after priming. These gels are given on a daily basis. This rhythm implies than for some women not responding to a first gel, priming can last up to three days, lengthening hospital stay and leading to maternal weariness. Maternal satisfaction during induction of labor is seldom analyzed. An intensification in gel administration implies a change in maternal management during the induction process, with shortened periods of rest between two gels and nearer periods of pain and discomfort, albeit on a theoretically shorter period. The way patients deal with this new rhythm compared to the classical in part of the evaluation in this study. All patients having a singleton pregnancy and an indication for term (≥ 37 weeks gestation age) induction with an unfavorable cervix and no contraindication to vaginal delivery will be eligible. Patients with fetuses in breech presentation, a scarred uterus, under 18 years, bearing a fetus with antenatally known malformation, not fluent in French or presenting an allergy to prostaglandins will be excluded. A written informed consent will be required before inclusion. The primary outcome will be the duration between first priming with prostaglandin gel and delivery. Secondary outcomes will be the satisfaction of patients with their induction process (measured through a survey answered during the in-hospital post-partum stay), the rate of cesarean section, the rate of hypertonia/hypercinesia during priming and induction requiring medical intervention, the length of active phase of labor (after 5 cm of dilation), the oxytocin doses used during delivery for induction or augmentation, initial neonatal (Apgar score, arterial cord pH and lactates, resuscitation maneuvers, transfer to intensive care unit) and maternal (post-partum hemorrhage, hyperthermia during labor, perineal laceration > 2nd degree and endometritis) morbidity and length of total hospital stay. The investigators calculated that a sample of 268 patients (134 in each group) will be necessary to detect a 30% reduction in duration between first priming and delivery in the experimental group (one gel every 12h) compared with the classical group. Mean time frame between first priming and delivery has been measured in our department in 2018 to 31.8 hours (standard deviation 27.6 hours).

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years
* Gestational age ≥ 37 weeks
* With indicated induction of labor and initial Bishop score under 6
* Without any contraindication to vaginal delivery
* Who consent to participate to the clinical research
* With French Medical Public Insurance

Exclusion Criteria:

* Multiple pregnancy
* Previous uterine scar (for myomas or cesarean section)
* Fetus not in cephalic presentation
* Allergy to prostaglandins
* Who not consent to participate to the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 268 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Time between gel administration and delivery | At inclusion (Day 0)
  Time between first gel administration for cervical priming and delivery
Time between gel administration and delivery | At 12 hours or 24 hours (after each gel administration)
  Change between cervical priming and delivery
Time between gel administration and delivery | Time 0 after the childbirth
  Time between first gel administration for cervical priming and delivery
Time between gel administration and delivery | Until 5 days postpartum (during in-hospital postpartum period)
  Time between first gel administration for cervical priming and delivery

SECONDARY OUTCOMES:
Maternal satisfaction | Until 5 days postpartum
  maternal satisfaction measured by survey self-administered during postpartum hospital stay
Cesarean section rate | During labor
Hypertonia / hypercinesia rate | During priming and induction
  Hypertonia (rise of uterus tone more than 10 minutes)/hypercinesia (more than 5 uterine contractions per 10 minutes) rate during priming and induction
Oxytocin dose during labor | During labor
  Induction or augmentation of Oxytocin doses
Length of active first phase of labor | During labor
  Induction or augmentation of active first phase of labor
Maternal morbidity | During labor
  Fever during labor, perineal laceration superior to 2nd degree, postpartum hemorrhage, endometritis
Neonatal immediate morbidity | 5 minutes after childbirth
  Assess if Apgar score is less than 7
Neonatal immediate morbidity | 5 minutes after childbirth
  Assess of arterial cord pH level
Neonatal immediate morbidity | 5 minutes after childbirth
  Assess of arterial cord lactate level
Neonatal immediate morbidity | 5 minutes after childbirth
  Concentration of arterial cord lactates level (in Mmol/L)
Neonatal immediate morbidity | 5 minutes after childbirth
  Occurence or not of resuscitation maneuvers in delivery room
Neonatal immediate morbidity | 5 minutes after childbirth
  Occurence or no transfer of the child to neonatal intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc VOLUMENIE, Principal Investigator — University Hospital of Martinique
Locations (1):
- University Hospital of Martinique, Fort-de-France, Martinique